CLINICAL TRIAL: NCT00730600
Title: Acute Changes in Biochemical Markers of Bone Resorption and Formation After THAI Traditional Massage
Brief Title: Effect of THAI Traditional Massage on Bone Markers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mahidol University (Other)
Responsible Party: Sunee - Saetung, Ramathibodi Hospital, Mahidol University, Bangkok, Thailand 10400
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: ID 02-50-30
Record Dates: First submitted 2008-08-06; First posted 2008-08-08 (Estimated); Last update posted 2008-08-08 (Estimated); Status verified 2008-07

CONDITIONS: Osteoporosis
Keywords: Thai Traditional massage; Bone Formation; Bone Resorption
MeSH Terms: conditions — Osteoporosis; Bone Resorption | interventions — Medicine, Thai Traditional

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): 1= THAI traditional massage
  Interventions: Procedure: Thai Traditional massage

INTERVENTIONS:
Procedure: Thai Traditional massage — Thai traditional massage for 2 hours by a single masseuse.
  Other Names: Thai massagae

SUMMARY:
The purpose of this study is to explore the skeletal effect of Thai traditional massage by examining the changes in biochemical markers of bone turnover immediately after the massage.

DETAILED DESCRIPTION:
Each subject received Thai traditional massage for 2 hours by a single masseuse.

ELIGIBILITY:
Inclusion Criteria:

* Healthy Thai women aged 20 to 40 years
* Have been massaged by Thai Traditional massage style

Exclusion Criteria:

* Hyperparathyroidism, Thyrotoxicosis, Diabetes Mellitus, Rheumatoid Arthritis, Cancer
* Antiresorptive agent, Teriparatide and Glucocorticoid
* Swelling Joints

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2007-06; Primary Completion 2007-09 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
Biochemical markers of bone resorption; C-terminal telopeptide of type I collagen (CTx-I) and of bone formation; total procollagen type 1 amino-terminal propeptide (P1NP)level | 2 hour

CONTACTS AND LOCATIONS:
Overall Officials: Sunee - Saetung, Msc, Principal Investigator — Ramathibodi Hospital, Mahidol University, Bangkok, Thailand 10400
Locations (1):
- Ramathibodi Hospital, Bangkok, Bangkok, Thailand